CLINICAL TRIAL: NCT02824536
Title: A Phase 1 Study of the Safety and Pharmacokinetics of the Combination of 3BNC117 and 10-1074 in HIV-uninfected Adults
Brief Title: 3BNC117 and 10-1074 in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YCO-0899
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: 3BNC117; 10-1074; Broadly neutralizing antibody; HIV Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — 3BNC117 antibody; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Participants will be randomized in a 3:1 ratio to receive one intravenous infusion of 3BNC117 and one intravenous infusion of 10-1074, each dosed at 10 mg/kg OR placebo (sterile saline), on day 0.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Drug: Placebo
- Group 2 (Experimental): Participants will be randomized in a 3:1 ratio to receive three intravenous infusions of 3BNC117 and three intravenous infusions of 10-1074, each dosed at 3 mg/kg OR placebo (sterile saline), on day 0, week 8, and week 16.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Drug: Placebo
- Group 3 (Experimental): Participants will be randomized in a 3:1 ratio to receive three intravenous infusions of 3BNC117 and three intravenous infusions of 10-1074, each dosed at 10 mg/kg OR placebo (sterile saline), on day 0, week 8, and week 16.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Drug: Placebo

INTERVENTIONS:
Drug: 3BNC117 — Intravenous Infusion of 3BNC117
  Other Names: Monoclonal Antibody 3BNC117
Drug: 10-1074 — Intravenous Infusion of 10-1074
  Other Names: Monoclonal Antibody 10-1074
Drug: Placebo — Intravenous Infusion of Sterile Saline (NaCl 0.9%)
  Other Names: Sterile Saline (NaCl 0.9%)

SUMMARY:
This is a phase 1 clinical trial to evaluate the safety and pharmacokinetics of the highly neutralizing anti-human immunodeficiency virus-1 monoclonal antibodies 3BNC117 and 10-1074, when given in combination, in human immunodeficiency virus (HIV)-uninfected individuals. This study is intended to support the development of the combination of 3BNC117 and 10-1074 mAbs for use as prophylaxis against HIV infection in healthy HIV-uninfected individuals at risk for HIV infection.

DETAILED DESCRIPTION:
The study will be conducted under a placebo-controlled, double blind, randomized allocation of the study products. Study participants in each study group will be randomized to receive intravenous infusions of 3BNC117 and 10-1074 or placebo. 3BNC117 and 10-1074 will be administered at 2 dose levels (3 mg/kg and 10 mg/kg). These doses were selected based on the planned development of subcutaneous formulations for the prophylactic use of these products. The study will consist of 3 groups. Enrollment in Group 1 will begin first and participants will be enrolled at least one day apart. Eight participants will be enrolled in each group; 6 will be randomized receive the study drugs and 2 will be randomized to receive placebo. Participants in Group 1 will receive a single infusion of each antibody at 10mg/kg at Week 0. Enrollment in Group 2 will begin only after Day 28 safety data from all participants in Group 1, including ophthalmologic exams, are available. Enrollment in Group 3 will begin only after the Day 28 safety data from all participants in Group 2 is available. If > 1 grade 3 or higher adverse events deemed probably or definitely related to the study drugs occurs in a single group, the next group will not be enrolled pending safety monitoring committee (SMC) review. Participants in Groups 2 and 3 will receive 3 infusions of each antibody at Weeks 0, 8, and 16, at a dose of either 3mg/kg or 10mg/kg. The antibodies will be administered sequentially via intravenous infusion. Each antibody will be administered over 60 minutes.

Following product infusions, study participants will return for safety assessments at multiple time points. Blood samples will be collected for safety testing at weeks 1, 2, and 4 following each infusion, then at multiple time points until the end of study follow up.

Baseline pharmacokinetic (PK) assessments will be performed before the start of the first infusion. Peak PK sampling for 3BNC117 will occur following the completion of the 3BNC117 infusion prior to the start of the 10-1074 infusion. Peak PK sampling for 10-1074 will occur following the completion of the 10-1074 infusion. Additional PK assessments will occur at multiple time points during study follow up. Study participants will be followed for a total of 24 weeks following the final antibody infusion.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 65.
* Amenable to HIV risk reduction counseling and agrees to maintain behavior consistent with low risk of HIV exposure.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) for the duration of the study.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection.
* History of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases) that in the opinion of the investigator would preclude participation.
* Within the 12 months prior to enrollment, the participant has a history of sexually transmitted infection.
* Chronic Hepatitis B or Hepatitis C infection.
* Laboratory abnormalities in the parameters listed:
* Absolute neutrophil count ≤ 2,000;
* Hemoglobin ≤ 12 gm/dL if female; ≤ 13.5 gm/dL if male;
* Platelet count ≤ 125,000;
* Alanine Aminotransferase (ALT) ≥ 1.25 x ULN; Aspartate Aminotransferase (AST) ≥ 1.25 x ULN;
* Alkaline phosphatase ≥ 1.5 x ULN
* Total bilirubin > 1.0 x ULN;
* Creatinine ≥1.1 x ULN;
* Pregnancy or lactation.
* Any vaccination within 14 days prior to infusion
* Receipt of any experimental HIV vaccine in the past.
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
The number of participants who experience adverse events within 1 week after the combination of 3BNC117 and 10-1074 infusion in all study groups. | 1 week following each combination of 3BNC117 and 10-1074 infusion
  Adverse events include signs, symptoms and laboratory abnormalities, in addition to local and systemic reactogenicity adverse events.

SECONDARY OUTCOMES:
Number of participants with induced anti-3BNC117 and anti-10-1074 antibodies | 8 weeks following each combination of 3BNC117 and 10-1074 infusion
Level of induced anti-3BNC117 and anti-10-1074 antibodies | 8 weeks following each combination of 3BNC117 and 10-1074 infusion
The number of participants who experience adverse events that occur during study follow up after 3BNC117 and 10-1074 infusions in all study groups. | 24-40 weeks
  Adverse events include signs, symptoms and laboratory abnormalities.

OTHER OUTCOMES:
Neutralization activity of serum from study participants against a panel of viruses as measured by the TZM.bl neutralization assay. | 24-40 weeks
Elimination half-life (t1/2) of 3BNC117 and 10-1074 | 24-40 weeks
Clearance (CL/F) of 3BNC117 and 10-1074 | 24-40 weeks
Volume of distribution (Vz/F) of 3BNC117 and 10-1074 | 24-40 weeks
Area under the plasma concentration versus time curve (AUC) of 3BNC117 and 10-1074 | 24-40 weeks
Decay Curve of of 3BNC117 and 10-1074 | 24-40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Cohen, MD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valente PK, Wu Y, Cohen YZ, Caskey M, Meyers K. Behavioral and social science research to support development of educational materials for clinical trials of broadly neutralizing antibodies for HIV treatment and prevention. Clin Trials. 2021 Feb;18(1):17-27. doi: 10.1177/1740774520948042. Epub 2020 Aug 24. PMID 32838558
- [Derived] Cohen YZ, Butler AL, Millard K, Witmer-Pack M, Levin R, Unson-O'Brien C, Patel R, Shimeliovich I, Lorenzi JCC, Horowitz J, Walsh SR, Lin S, Weiner JA, Tse A, Sato A, Bennett C, Mayer B, Seaton KE, Yates NL, Baden LR, deCamp AC, Ackerman ME, Seaman MS, Tomaras GD, Nussenzweig MC, Caskey M. Safety, pharmacokinetics, and immunogenicity of the combination of the broadly neutralizing anti-HIV-1 antibodies 3BNC117 and 10-1074 in healthy adults: A randomized, phase 1 study. PLoS One. 2019 Aug 8;14(8):e0219142. doi: 10.1371/journal.pone.0219142. eCollection 2019. PMID 31393868